CLINICAL TRIAL: NCT02598999
Title: Randomized, Double Blind, Placebo-controlled Study of the Safety, Tolerability and Pharmacokinetics After Single Ascending Doses or Multiple Ascending Doses of OSCN-, bLF or ALX-009 in Healthy Male and CF and Non-CF Bronchiectasis Patients
Brief Title: Dose Escalation Study of ALX-009 in Healthy Men and Cystic Fibrosis (CF) and Non-CF Bronchiectasis Patients
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Financial issues
Sponsor: Alaxia SAS (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ALX-009-CL-038; 2014-002401-38 (EudraCT Number)
Record Dates: First submitted 2015-11-04; First posted 2015-11-06 (Estimated); Last update posted 2022-02-03 (Actual); Status verified 2022-01

CONDITIONS: Cystic Fibrosis; Bronchiectasis
MeSH Terms: conditions — Cystic Fibrosis; Bronchiectasis | interventions — hypothiocyanite ion

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Part I, SAD (Experimental): Single administration of OSCN- or bLF or Placebo in healthy male volunteers
  Interventions: Drug: OSCN-; Drug: bLF; Drug: Placebo
- Part II, SAD and MAD (Experimental): Single and multiple administrations of ALX-009 or Placebo in healthy male volunteers
  Interventions: Drug: ALX-009; Drug: Placebo
- Part III, MAD (Experimental): Multiple administrations of OSCN- or bLF or Placebo in CF patients in healthy volunteers
  Interventions: Drug: OSCN-; Drug: bLF; Drug: Placebo
- Part IV, MAD (Experimental): Multiple administrations of ALX-009 or Placebo in healthy volunteers and in patients (CF and NCFBE)
  Interventions: Drug: ALX-009; Drug: Placebo

INTERVENTIONS:
Drug: ALX-009 — Solution for inhalation administered through nebulization
  Other Names: Association of OSCN- and bLF
  Arms: Part II, SAD and MAD; Part IV, MAD
Drug: OSCN- — Solution for inhalation administered through nebulization
  Other Names: Hypothiocyanite
  Arms: Part I, SAD; Part III, MAD
Drug: bLF — Solution for inhalation administered through nebulization
  Other Names: bovine Lactoferrin
  Arms: Part I, SAD; Part III, MAD
Drug: Placebo — Solution for inhalation administered through nebulization, Sodium Chloride 0.9%

SUMMARY:
This is a Phase 1, randomized, double-blind, placebo-controlled study to evaluate the safety, tolerability and pharmacokinetics of a single ascending doses (SAD) and multiple ascending doses (MAD) of Hypothiocyanite (OSCN-), bovine lactoferrin (bLF) and their combination (ALX-009) in healthy male volunteers and patients suffering from cystic fibrosis (CF) and non-CF bronchiectasis (NCFBE).

DETAILED DESCRIPTION:
Part I: SAD of OSCN- and bLF in healthy male volunteers (cohorts 1 to 3) - Part II: SAD and MAD of ALX-009 in healthy male volunteers (cohorts 4 and 5) - Part III: MAD of OSCN- and bLF in patients suffering from cystic fibrosis (cohort III-1) and in healthy volunteers (cohorts III-2 and III-3) - Part IV: MAD of ALX-009 in healthy volunteers (Part IVa - Cohorts IV-1a to IV-3a) and in patients (Part IVb - Cohorts IV-1b to IV-3b)

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subject or
* Patient suffering from cystic fibrosis defined as a positive sweat chloride test or CF-causing mutations, documented in the patient's medical record or patient suffering from non-CF and non COPD bronchiectasis with a diagnosis confirmed by a chest CT scan demonstrating bronchiectasis in 1 or more lobes documented in the patient's medical record
* Aged between 18 and 50 years inclusive
* Subject's Body Mass Index between 18 and 30 kg/m²
* Subject with normal blood pressure, heart rate, ECG recording and laboratory parameters at the screening visit
* Subject having given a written informed consent prior to selection
* Subject covered by Health Insurance System and/ or in compliance with the recommendations of National Law in force relating to biomedical research

Specific Inclusion Criteria for patients:

* FEV1 more than or equal to 60% of predicted normal value
* Subject in a stable state (no exacerbation for 1 month or prescription of antibiotic by intravenous route)
* Females of childbearing potential: commitment to consistently and correctly use an acceptable method of birth control for the duration of the trial and for 4 months after the last study drug administration / Female of non-childbearing potential: either surgically sterilized or at least 1 year postmenopausal

Exclusion Criteria:

* Presence of cardiovascular, pulmonary, gastro-intestinal, hepatic, renal, metabolic, haematological, neurologic, psychiatric, systemic or infectious disease
* Frequent headaches and/or migraines, recurrent nausea and/or vomiting
* Symptomatic hypotension
* Blood donation (including in the frame of a clinical trial) within 2 months before administration
* General anaesthesia within 3 months before administration
* Presence or history of drug hypersensitivity, or any allergic disease
* Medical history of reactions to cow's milk proteins
* Subject who can not be contacted in case of emergency
* History or presence of drug or alcohol abuse
* Positive Hepatitis B surface (HBs) antigen or anti Hepatitis C virus (HCV) antibody, or positive results for Human Immunodeficiency Virus (HIV) 1 or 2 tests
* Subject who, in the judgement of the Investigator, is likely to be non-compliant or uncooperative during the study, or unable to cooperate because of a language problem, poor mental development.

Specific exclusion criteria for study Parts III and IV:

* Known bronchial hyper-reactivity to drug inhalation
* Known contra-indication to inhaled salbutamol
* Subject with bronchial hyper-reactivity, defined by a positive response to bronchodilator with FEV1 increase ≥ 200 mL

Specific exclusion crtieria for patients:

* Active allergic bronchopulmonary aspergillosis currently treated
* Medical history of allergic bronchopulmonary aspergillosis in the past 2 years.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 92 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2021-12 (Actual); Study Completion 2021-12 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability: number of subjects who experience serious adverse events, adverse events, potential clinically significant changes in ECG, 24-holter, vital signs, physical examinations, laboratory tests, spirometry, O2 saturation (Part III only) | Day (D) 8 post dosing for part I and D14 post dosing for parts II, III and IV

SECONDARY OUTCOMES:
Maximal concentration (Cmax) of bLF and SCN- in plasma, sputum and urine (for SCN- only) | D8 post dosing for part I and D14 post dosing for parts II, III and IV
Area under the curve (AUC) of bLF and SCN- in plasma, sputum and urine (for SCN- only) | D8 post dosing for part I and D14 post dosing for parts II, III and IV
First time to reach Cmax (Tmax) of bLF and SCN- in plasma, sputum and urine (for SCN- only) | D8 post dosing for part I and D14 post dosing for parts II, III and IV
Concentration half life of bLF and SCN- in plasma, sputum and urine (for SCN- only) | D8 post dosing for part I and D14 post dosing for parts II, III and IV
Concentration of anti-bLF antibodies in blood and sputum | D8 post dosing for part I and D14 post dosing for parts II, III and IV
Concentration of IL-1β in blood and sputum | D8 post dosing for part I and D14 post dosing for parts II, III and IV
Concentration of IL-6 in blood and sputum | D8 post dosing for part I and D14 post dosing for parts II, III and IV
Concentration of IL-8 in blood and sputum | D8 post dosing for part I and D14 post dosing for parts II, III and IV
Concentration of IL-10 in blood and sputum | D8 post dosing for part I and D14 post dosing for parts II, III and IV
Concentration of TNF-α in blood and sputum | D8 post dosing for part I and D14 post dosing for parts II, III and IV
Concentration of SC5b-9 in blood | D8 post dosing for part I and D14 post dosing for parts II, III and IV
Concentration of total IgE in blood | D8 post dosing for part I and D14 post dosing for parts II, III and IV
For patients only, quantitative assessment of different species in sputum | D7 post dosing
  Staphylococcus aureus, Staphylococcus aureus MRSA, Pseudomonas aeruginosa, Pseudomonas aeruginosa MDR, Haemophilus influenzae, Stenotrophomonas maltophilia, Achromobacter xylosoxidans, Burkholderia cepacia complex, Aspergillus fumigatus and Aspergillus terreus
For patients only, volume of sputum over 24hours period | D8 post dosing

OTHER OUTCOMES:
For patients only, characterization of sputum microbiota using genomic technologies | D14 post dosing

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle Durieu, Prof., MD, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Eurofins Optimed, Grenoble, France